CLINICAL TRIAL: NCT04439838
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 1595043 (Single-blind, Partially Randomised, Placebo-controlled, Parallel (Sequential) Group Design) in Healthy Male Subjects
Brief Title: A Study in Healthy Men to Test How Different Doses of BI 1595043 Are Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1445-0001; 2020-001036-10 (EudraCT Number)
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Results first posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- 1 mg BI 1595043 (Experimental): 1 mg BI 1595043
  Interventions: Drug: BI 1595043
- 3 mg BI 1595043 (Experimental): 3 mg BI 1595043
  Interventions: Drug: BI 1595043
- 6 mg BI 1595043 (Experimental): 6 mg BI 1595043
  Interventions: Drug: BI 1595043
- 12 mg BI 1595043 (Experimental): 12 mg BI 1595043
  Interventions: Drug: BI 1595043
- 25 mg BI 1595043 (Experimental): 25 mg BI 1595043
  Interventions: Drug: BI 1595043
- 50 mg BI 1595043 (Experimental): 50 mg BI 1595043
  Interventions: Drug: BI 1595043
- 90 mg BI 1595043 (Experimental): 90 mg BI 1595043
  Interventions: Drug: BI 1595043
- 160 mg BI 1595043 (Experimental): 160 mg BI 1595043
  Interventions: Drug: BI 1595043
- Matching Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1595043 — BI 1595043
  Arms: 1 mg BI 1595043; 12 mg BI 1595043; 160 mg BI 1595043; 25 mg BI 1595043; 3 mg BI 1595043; 50 mg BI 1595043; 6 mg BI 1595043; 90 mg BI 1595043
Drug: Placebo — Placebo
  Arms: Matching Placebo

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability and pharmacokinetics (PK) of BI 1595043 in healthy male subjects following oral administration of single rising doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* BMI of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation
* Male subjects who meet any of the following criteria from at least 30 days before the first administration of trial medication until 30 days after trial completion:

  * Use of adequate contraception, e.g. use of condom (male subjects) plus any of the following methods (female partners): intrauterine device, hormonal contraception (e.g. implants, injectables, combined oral or vaginal contraceptives) that started at least 2 months prior to first drug administration to the male subject, or barrier method (e.g. diaphragm with spermicide), or surgically sterilised (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy), or postmenopausal, defined as at least 1 year of spontaneous amenorrhea
  * Sexually abstinent
  * Vasectomised (vasectomy at least 1 year prior to enrolment) in combination with a barrier method (e.g. condom)
* Unprotected sexual intercourse with a pregnant female partner and sperm donation is not allowed throughout the study and until 30 days after trial completion

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A single-blind, partially randomised, placebo-controlled study to test how different doses of BI 1595043 are tolerated in healthy men.
Pre-assignment Details: Only subjects that met all the inclusion and none of the exclusion criteria were to be entered in the study. All subjects were free to withdraw from the clinical trial at any time for any reason given. Close monitoring was adhered throughout the trial conduct.
Groups:
- Matching Placebo: Matching placebo administered as single oral dose with 240 milliliter (mL) of water after an overnight fast of at least 10 hours.
- 1 mg BI 1595043: Participants were administered 0.4 ml oral solution of BI 1595043 concentrated 2.5 milligram (mg)/ milliliter (mL) (total dose: 1 mg BI 1595043) as single dose once daily with 240 mL of water after an overnight fast of at least 10 hours.
- 3 mg BI 1595043: Participants were administered 1.2 ml oral solution of BI 1595043 concentrated 2.5 mg/mL (total dose: 3 mg BI 1595043) as single dose once daily with 240 mL of water after an overnight fast of at least 10 hours.
- 6 mg BI 1595043: Participants were administered 2.4 ml oral solution of BI 1595043 concentrated 2.5 mg/mL (total dose: 6 mg BI 1595043) as single dose once daily with 240 mL of water after an overnight fast of at least 10 hours.
- 12 mg BI 1595043: Participants were administered 4.8 ml oral solution of BI 1595043 concentrated 2.5 mg/mL (total dose: 12 mg BI 1595043) as single dose once daily with 240 mL of water after an overnight fast of at least 10 hours.
- 25 mg BI 1595043: Participants were administered 10 ml oral solution of BI 1595043 concentrated 2.5 mg/mL (total dose: 25 mg BI 1595043) as single dose once daily with 240 mL of water after an overnight fast of at least 10 hours.
- 50 mg BI 1595043: Participants were administered 20 ml oral solution of BI 1595043 concentrated 2.5 mg/mL (total dose: 50 mg BI 1595043) as single dose once daily with 240 mL of water after an overnight fast of at least 10 hours.
- 90 mg BI 1595043: Participants were administered 36 ml oral solution of BI 1595043 concentrated 2.5 mg/mL (total dose: 90 mg BI 1595043) as single dose once daily with 240 mL of water after an overnight fast of at least 10 hours.
- 160 mg BI 1595043: Participants were administered 64 ml oral solution of BI 1595043 concentrated 2.5 mg/mL (total dose: 160 mg BI 1595043) as single dose once daily with 240 mL of water after an overnight fast of at least 10 hours.
Period: Overall Study
Arm/Group | Matching Placebo | 1 mg BI 1595043 | 3 mg BI 1595043 | 6 mg BI 1595043 | 12 mg BI 1595043 | 25 mg BI 1595043 | 50 mg BI 1595043 | 90 mg BI 1595043 | 160 mg BI 1595043
Started | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed (planned observation time) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The TS included all subjects who were randomised and treated with at least 1 dose of trial drug. The treatment assignment was determined based on the first treatment the subjects received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Matching Placebo | 1 mg BI 1595043 | 3 mg BI 1595043 | 6 mg BI 1595043 | 12 mg BI 1595043 | 25 mg BI 1595043 | 50 mg BI 1595043 | 90 mg BI 1595043 | 160 mg BI 1595043 | Total
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] — Treated Set (TS).
  Years | 34.3 (8.1) | 39.8 (4.3) | 37.8 (8.6) | 40.2 (4.8) | 35.3 (9.1) | 34.2 (11.1) | 29.0 (4.0) | 37.7 (8.7) | 34.2 (10.0) | 35.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Treated Set (TS).
  Participants
    Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Male | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Treated Set (TS).
  Participants
    Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
    Not Hispanic or Latino | 15 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 62
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Treated Set (TS).
  Participants
    American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    White | 14 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 4 | 59
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Drug-related Adverse Events (AEs)
Description: Percentage of participants with drug-related adverse events (AEs) is reported.
Time Frame: From drug administration until end of trial, up to 15 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Matching Placebo | 1 mg BI 1595043 | 3 mg BI 1595043 | 6 mg BI 1595043 | 12 mg BI 1595043 | 25 mg BI 1595043 | 50 mg BI 1595043 | 90 mg BI 1595043 | 160 mg BI 1595043
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Percentage of participants | 12.5 | 0.0 | 16.7 | 0.0 | 0.0 | 16.7 | 16.7 | 0.0 | 0.0

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 1595043 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-inf)
Description: Area under the concentration-time curve of BI 1595043 in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf) is reported.
Time Frame: Within 3 hours prior to drug administration and 0.5, 1, 1.5, 2*, 2.5, 3, 4, 6, 8, 10, 12, 24, 34, 48, 72, 96, 120, 144, 168 and 192 hours after drug administration. * Only for dose group "12 mg BI 1595043".
Population: Pharmacokinetic parameter analysis set (PKS): This set included all subjects in the treated set (TS) who provided at least 1 pharmacokinetic (PK) endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS, even if he contributed only 1 PK parameter value for 1 period to the statistical assessment. Only participants with non-missing values are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours * nanomole / Liter
Arm/Group | 1 mg BI 1595043 | 3 mg BI 1595043 | 6 mg BI 1595043 | 12 mg BI 1595043 | 25 mg BI 1595043 | 50 mg BI 1595043 | 90 mg BI 1595043 | 160 mg BI 1595043
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5
Hours * nanomole / Liter | 294 (26.9) | 571 (14.9) | 958 (19.9) | 1850 (19.6) | 3210 (19.7) | 5510 (20.3) | 12300 (11.8) | 18700 (10.1)

3. Secondary Outcome: Maximum Measured Concentration of BI 1595043 in Plasma (Cmax)
Description: Maximum measured concentration of BI 1595043 in plasma (Cmax) is reported.
Time Frame: as for outcome 2
Population: Pharmacokinetic parameter analysis set (PKS): This set included all subjects in the treated set (TS) who provided at least 1 pharmacokinetic (PK) endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS, even if he contributed only 1 PK parameter value for 1 period to the statistical assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole / Liter
Arm/Group | 1 mg BI 1595043 | 3 mg BI 1595043 | 6 mg BI 1595043 | 12 mg BI 1595043 | 25 mg BI 1595043 | 50 mg BI 1595043 | 90 mg BI 1595043 | 160 mg BI 1595043
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Nanomole / Liter | 23.6 (16.7) | 78.4 (10.9) | 119 (21.2) | 286 (20.5) | 516 (26.2) | 1100 (27.1) | 2500 (20.0) | 4620 (21.8)

ADVERSE EVENTS:
Time Frame: From drug administration until end of trial, up to 15 days.
Description: Treated Set (TS): The TS included all subjects who were randomised and treated with at least 1 dose of trial drug. The treatment assignment was determined based on the first treatment the subjects received.
Arm/Group | Matching Placebo | 1 mg BI 1595043 | 3 mg BI 1595043 | 6 mg BI 1595043 | 12 mg BI 1595043 | 25 mg BI 1595043 | 50 mg BI 1595043 | 90 mg BI 1595043 | 160 mg BI 1595043
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/16 | 0/6 | 1/6 | 1/6 | 2/6 | 3/6 | 4/6 | 0/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Matching Placebo (N=16) | 1 mg BI 1595043 (N=6) | 3 mg BI 1595043 (N=6) | 6 mg BI 1595043 (N=6) | 12 mg BI 1595043 (N=6) | 25 mg BI 1595043 (N=6) | 50 mg BI 1595043 (N=6) | 90 mg BI 1595043 (N=6) | 160 mg BI 1595043 (N=6)
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angular cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT04439838/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT04439838/SAP_001.pdf